CLINICAL TRIAL: NCT02958566
Title: Multimodal Narcotic Limited Perioperative Pain Control With Colorectal Surgery as Part of an Enhanced Recovery After Surgery Protocol: A Randomized Prospective Single- Center Trial.
Brief Title: Multimodal Narcotic Limited Perioperative Pain Control With Colorectal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois College of Medicine at Peoria (Other)
Responsible Party: Principal Investigator, Steven Tsoraides, Assistant Professor of Clinical Surgery, OSF Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 825977-4
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Colon Cancer; Colon Diverticulosis; Colonic Neoplasms; Colonic Diverticulitis; Pain, Postoperative; Ileus; Ileus Paralytic; Ileus; Mechanical; Constipation Drug Induced; Constipation; Rectum Cancer; Rectum Neoplasm
Keywords: Pain control; Post-operative pain; Narcotic; Non-narcotic; Side effect; Toxicity
MeSH Terms: conditions — Colonic Neoplasms; Diverticulosis, Colonic; Diverticulitis, Colonic; Pain, Postoperative; Ileus; Constipation; Rectal Neoplasms; Agnosia | interventions — Acetaminophen; Gabapentin; Orphenadrine; Lidocaine; Bupivacaine; Ketamine; Methadone; Tramadol; Ketorolac; Ketorolac Tromethamine; Morphine; Fentanyl; Hydromorphone; oxycodone-acetaminophen; Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Narcotic (Active Comparator): Morphine, Dilaudid or Fentanyl patient controlled anesthesia (PCA) for the immediate postoperative period, in addition to Norco 5-325 mg 1-2 tabs Q4H PRN, or equivalent medication.
  Post-operative day 1: PCA will be discontinued and the patients will have IV narcotics PRN: Morphine 1-2 mg Q2H PRN, fentanyl 50-75 mcg Q2H PRN or Dilaudid 0.5 mg Q2H PRN
  Interventions: Drug: Morphine Sulfate; Drug: Fentanyl; Drug: Dilaudid; Drug: HYDROCODONE/ACETAMINOPHEN 5 Mg-325 Mg ORAL TABLET
- Non-Narcotic (Experimental): Gabapentin 300 mg PO, orphenadrine 60 mg IV, acetaminophen 1000 mg PO or IV on Morning of surgery. Lidocaine 100 mg prior to incision, lidocaine 1mg/kg/hour during procedure, marcaine in all incisions. Ketamine and methadone per anesthesia. Acetaminophen 1000 mg PO or IV, gabapentin 300 mg PO, tramadol 50 mg PO in PACU. Acetaminophen 600 mg PO Q 6 hours, tramadol 50 mg PO Q 6 hours, gabapentin 300 mg PO Q 6 hours, orphenadrine 60 mg IV Q 12 hours, ketorolac 15 mg IV Q 6 hours for 48 hours post-operatively.
  Interventions: Drug: Acetaminophen; Drug: Gabapentin; Drug: Orphenadrine; Drug: Lidocaine; Drug: Marcaine; Drug: Ketamine; Drug: Methadone; Drug: Tramadol; Drug: Ketorolac; Drug: Morphine Sulfate; Drug: Fentanyl; Drug: Dilaudid; Drug: Hydrocodone-Acetaminophen Tab 5-325 MG

INTERVENTIONS:
Drug: Acetaminophen
  Other Names: Tylenol; Ofirmev
  Arms: Non-Narcotic
Drug: Gabapentin
  Other Names: Neurontin
  Arms: Non-Narcotic
Drug: Orphenadrine
  Other Names: Norflex
  Arms: Non-Narcotic
Drug: Lidocaine
  Arms: Non-Narcotic
Drug: Marcaine
  Arms: Non-Narcotic
Drug: Ketamine
  Arms: Non-Narcotic
Drug: Methadone
  Arms: Non-Narcotic
Drug: Tramadol
  Other Names: Ultram
  Arms: Non-Narcotic
Drug: Ketorolac
  Other Names: Toradol
  Arms: Non-Narcotic
Drug: Morphine Sulfate
  Arms: Non-Narcotic
Drug: Fentanyl
  Arms: Non-Narcotic
Drug: Dilaudid
  Arms: Non-Narcotic
Drug: Hydrocodone-Acetaminophen Tab 5-325 MG
  Other Names: Norco
  Arms: Non-Narcotic
Drug: Morphine Sulfate — PCA
  Arms: Narcotic
Drug: Fentanyl — PCA
  Arms: Narcotic
Drug: Dilaudid — PCA
  Arms: Narcotic
Drug: HYDROCODONE/ACETAMINOPHEN 5 Mg-325 Mg ORAL TABLET — Breakthrough
  Other Names: Norco
  Arms: Narcotic

SUMMARY:
The General Objective of this study is to investigate the cost and efficacy of treating patients undergoing colorectal surgical resections with an opioid limited pain control regimen as part of an Enhanced Recovery After Surgery (ERAS) Protocol. This group will be compared to a traditional opioid based pain control regimen.

DETAILED DESCRIPTION:
Postoperative ileus is a well-known problem for patients who have undergone a colorectal procedure. It is manifested as abdominal distension, accumulation of gas and fluid within the bowels and delayed bowel function (flatus or defecation). It is estimated that with traditional perioperative care for open colon resection postoperative ileus can lead to a length of stay (LOS) of 10 days. Such factors include the use of narcotics, immobilization, over-hydration with IV fluid etc. With about 350,000 colon and small bowel resections occurring annually and a bill to the healthcare system greater than US $20 billion, even decreasing LOS by one or two days can result in substantial cost savings.

All patients undergoing colorectal surgery require medications for pain control. The mainstay of current treatment includes narcotics/opioids. The effect of these medicines on mu receptors of the intestine contribute to delayed bowel function. Protocols that limit the use of narcotics/opioids may reduce the risk of ileus, thus reducing length of stay and reducing cost.

A prospective randomized clinical trial at a single tertiary referral academic affiliated medical center (OSF St. Francis Medical Center). Patients undergoing minimally invasive (laparoscopic or robotic) colorectal resection will be considered for inclusion. Surgery will be performed by two surgeons participating in the study protocol. Patient accrual is intended to begin May 1, 2016 and terminate either after 80 patients have been accrued or December 31, 2018, whichever is first. Informed consent will be obtained and preoperative education will be provided (appendix A). Patients will be randomized to one of two groups. The randomization scheme is a random-permuted-block design without stratification. The block size is a random number between 4 and 8. Personnel who are unassociated with patient screening, enrollment, or follow-up will create the allocation sequence and will use a computerized, random number generator. The allocation sequence will be transferred to sequentially numbered, opaque envelopes for purposes of allocation concealment. Clinical trial coordinators/physicians will verify patient eligibility and informed consent before opening the envelope to obtain the treatment assignment. The experimental group will be placed on a narcotic limited protocol as described below. All used medications are FDA approved. No investigational medicines will be used.

ELIGIBILITY:
Inclusion Criteria:

* Males or females above the age of 18
* Patients undergoing laparoscopic or robotic colorectal resections

Exclusion Criteria:

* History of constipation
* Pre-existing use of narcotics or opioids
* Pre-existing renal or hepatic failure
* Mental illness, mental retardation, or inability to participate in informed consent due to mental status
* Pre-existing dementia
* Allergy to any protocol medication
* Emergency operation
* Subjects who are incarcerated or wards of the state
* Minors
* Subjects with inflammatory bowel disease, active colitis, or pre-existing intra-abdominal inflammation. Diverticulitis without active infection/inflammation will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay | 30 days
  Total time in hospital from admission to discharge
Days to Return of Bowel Function | 30 days
  Time from operation to first passage of flatus or bowel movement
Medication cost | 30 days
  Total cost of inpatient medications
Hospital stay cost | 30 days
  Total cost of hospital stay

SECONDARY OUTCOMES:
Amount of narcotics used | 30 days
  Total amount of narcotics patient consumed
Complications | 30 days
  Death, prolonged ileus (insertion of NG tube or lack of bowel function on POD 3), respiratory failure, renal failure, SSI, leak, pneumonia, UTI, DVT/PE, cardiac event/MI
Mortality | 30 days
Patient satisfaction | 30 days
  Measured using a survey given to patient at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Steven S Tsoraides, MD, MPH, Principal Investigator — University of Illinois College of Medicine at Peoria
Locations (1):
- Uicomp, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Muller S, Zalunardo MP, Hubner M, Clavien PA, Demartines N; Zurich Fast Track Study Group. A fast-track program reduces complications and length of hospital stay after open colonic surgery. Gastroenterology. 2009 Mar;136(3):842-7. doi: 10.1053/j.gastro.2008.10.030. Epub 2008 Nov 1. PMID 19135997
- [Result] Serclova Z, Dytrych P, Marvan J, Nova K, Hankeova Z, Ryska O, Slegrova Z, Buresova L, Travnikova L, Antos F. Fast-track in open intestinal surgery: prospective randomized study (Clinical Trials Gov Identifier no. NCT00123456). Clin Nutr. 2009 Dec;28(6):618-24. doi: 10.1016/j.clnu.2009.05.009. Epub 2009 Jun 17. PMID 19535182
- [Result] Lubawski J, Saclarides T. Postoperative ileus: strategies for reduction. Ther Clin Risk Manag. 2008 Oct;4(5):913-7. doi: 10.2147/tcrm.s2390. PMID 19209273